CLINICAL TRIAL: NCT01936090
Title: Phase I/II Bortezomib, Melphalan and Low Dose TBI Conditioning for Patients Undergoing Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: Bortezomib, Melphalan, and Total-Body Irradiation Before Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1286; NCI-2013-01646 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Mod12-008546-08; MC1286 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Whole-Body Irradiation; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bortezomib, TBI, melphalan, stem cell transplant) (Experimental): Conditioning regimen: Patients receive bortezomib IV on days -5 and -2, TBI BID on days -5 and -2, and melphalan IV over 1 hour on days -4 and -3.
  Transplant: Patients undergo autologous bone marrow or peripheral blood stem cell transplant on day 0.
  Interventions: Drug: Bortezomib; Radiation: Total-Body Irradiation; Drug: Melphalan; Procedure: Autologous Bone Marrow Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bortezomib — Given IV
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole-Body Irradiation
Drug: Melphalan — Given IV
  Other Names: Alkeran
Procedure: Autologous Bone Marrow Transplantation — Undergo autologous bone marrow transplant
  Other Names: ABMT; Autologous Bone Marrow Transplant; Autologous Marrow Transplantation
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: Autologous Stem Cell Transplantation
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of bortezomib when given together with melphalan, and total-body irradiation before stem cell transplant and to see how well it works in treating patients with multiple myeloma. Giving chemotherapy and total-body irradiation before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. The stem cells that were collected from the patient's blood or bone marrow are returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and total-body irradiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of bortezomib that can be added to high dose melphalan and low dose total body irradiation as part of conditioning chemotherapy for myeloma. (Phase I) II. To determine the efficacy of the bortezomib added to high dose melphalan and low dose total-body irradiation (TBI) in patients with myeloma undergoing stem cell transplantation, as defined by achievement of complete response (CR). (Phase II)

SECONDARY OBJECTIVES:

I. To examine the toxicities associated with addition of bortezomib to high dose melphalan and TBI in patients with multiple myeloma (MM).

II. To determine the progression free rate at 1 and 2 years.

TERTIARY OBJECTIVES:

I. To determine the proportion of patients achieving a minimal residual disease (MRD) negative status.

II. To assess the HevyLite assay prior to and during treatment.

OUTLINE: This is a phase I, dose-escalation study of bortezomib followed by a phase II study.

CONDITIONING REGIMEN: Patients receive bortezomib intravenously (IV) on days -5 and -2, TBI twice daily (BID) on days -5 and -2, and melphalan IV over 1 hour on days -4 and -3.

TRANSPLANT: Patients undergo autologous bone marrow or peripheral blood stem cell transplant on day 0.

After completion of study treatment, patients are followed up at 100 days and then every 90 days for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine =< 2 mg/dL
* Serum total bilirubin =< 1.5 X upper limit of normal (ULN)
* Platelet count >= 30,000/μL
* Hemoglobin >= 8.0 g/dL
* Diagnosis of myeloma for which autologous stem cell transplant is being considered
* Measurable disease of multiple myeloma at the time of baseline values for disease assessment as defined by at least one of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Bone marrow plasma cells >= 30%
* NOTE:

  * For patients with no relapse prior to transplant, measurable disease at the time of diagnosis
  * For patients who have had a disease relapse prior to transplant, measurable disease at the time of the most recent relapse immediately prior to transplant.
  * If the patient had treatment for the relapsed disease prior to transplant, the patient must have measurable disease at the time of relapse prior to this therapy
* Patient is considered for autologous stem cell transplantation with full dose melphalan (200 mg/m^2)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Recovered from non-hematological toxicity of previous chemotherapy (excludes grade 1 neurotoxicity)
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Ejection fraction >= 45%
* Corrected pulmonary diffusion capacity of greater than or equal to 50%
* Forced expiratory volume in one second (FEV1) >= 50%
* Forced vital capacity (FVC) >= 50%
* Negative pregnancy test performed =< 14 days prior to registration, for women of childbearing potential only
* Willing to return to Mayo Clinic Rochester, for treatment and follow-up

  * Note: During the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide blood and bone marrow samples for correlative research purposes

Exclusion Criteria:

* Prior autologous or allogeneic bone marrow/peripheral blood stem cell transplant
* More than two prior regimens for therapy of MM
* Myocardial infarction within 6 months prior to enrollment, or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; NOTE: prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Seroreactivity for human immunodeficiency virus (HIV), human T-cell lymphotrophic virus (HTLV) I or II, hepatitis B virus (HBV), hepatitis C virus (HCV)
* Other active malignancy < 2 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix or low-risk prostate cancer after curative therapy

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Any of the following:

  * Pregnant women or women of reproductive capability who are unwilling to use effective contraception (2 effective methods of contraception, at the same time) from the time of signing the informed consent through 30 days after the last dose of study treatment, OR unwilling to agree to completely abstain from heterosexual intercourse
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 30 days after stopping treatment
  * Unwilling to agree to completely abstain from heterosexual intercourse
* Other co-morbidity, which would interfere with patient's ability to participate in the trial, e.g. uncontrolled infection, uncompensated lung disease or psychiatric illness
* Concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Known allergies to any of the components of the investigational treatment regimen or required ancillary treatments
* Patient has >= grade 2 peripheral neuropathy
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (phase I) | Day 36
The number and severity of all adverse events (phase I) | Up to 3 years
  Will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Proportion of complete responses (CR) defined as a CR noted as the objective status on two consecutive evaluations (phase II) | Up to 3 years
  Will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. 95% confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
CR rate at day 100 estimated by the total number of patients who achieve a complete CR by day 100 post-transplant divided by the total number of evaluable patients | At day 100
  Exact binomial 95% confidence intervals for the true CR rate at day 100 will be calculated.
Time to progression | Time from registration to the earliest date with documentation of disease progression, assessed at 1 year
  Will be estimated using the method of Kaplan-Meier.
Time to progression | Time from registration to the earliest date with documentation of disease progression, assessed at 2 years
  Will be estimated using the method of Kaplan-Meier.
Maximum grade for each type of adverse event | Up to 3 years
  Will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
Proportion of patients who achieve MRD negative status estimated by the number of patients who are MRD negative divided by the total number of evaluable patients who achieve a CR | Up to 3 years
  Exact binomial 95% confidence intervals for the true MRD negative rate will be calculated.
Abnormal ratio and suppressed uninvolved immunoglobulin assessed by HevyLite assay | Up to 3 years
  The correlation of these categories with whether MRD is present (yes vs. no) will be evaluated using Fisher's exact test. In addition, the relationship between these categories and time to progression will be evaluated using Kaplan-Meier methods and log-rank statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States